CLINICAL TRIAL: NCT03619148
Title: The Incidence and Severity of Upper Respiratory Tract Symptoms Associated With The Use of High-Flow Humidified Nasal Oxygen (HFNO)
Brief Title: The Incidence of Respiratory Symptoms Associated With the Use of HFNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS-233721; 18/LO/1133 (Other: Research Ethics Committee)
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 2 sub group will be recruited:
  1. patient undergoing TOE
  2. Staff volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Flow Humidified Nasal Oxygen - TOE participants (Other): High-Flow Humidified Nasal Oxygen - standard care
  Interventions: Device: High-Flow Humidified Nasal Oxygen
- High-Flow Humidified Nasal Oxygen (Active Comparator): High-Flow Humidified Nasal Oxygen - staff volunteers
  Interventions: Device: High-Flow Humidified Nasal Oxygen

INTERVENTIONS:
Device: High-Flow Humidified Nasal Oxygen — High-Flow Humidified Nasal Oxygen

SUMMARY:
Optiflow (high flow humified nasal oxygen) is used in several settings frequently (ICU, during elective general anaesthesia- commonly here on the TOE list, in certain ENT patients, and more commonly now in obese or obstetric patients for preoxygenation). To the investigators knowledge no one has quantified the common complications associated with it (based on a literature search in November 2017 using PubMed and Google; using the search terms "high flow nasal oxygen" combined with "complications", "side effects", "nasal dryness" and "epistaxis"). The investigators were unable to find any existing research that examined the days following HFNO use and specifically looked for minor side effects) The investigators have had anecdotal feedback from patients that they tend to experience respiratory symptoms post HFNO.

THe investigators would like to determine how often this occurs and how long it lasts for which would be pertinent to consent, and informing patients prior to the procedure, and also serve to improve the literature on this up and coming technique.

DETAILED DESCRIPTION:
The study aims to evaluate what is the frequency and severity of respiratory tract symptoms following the use of high flow nasal humidified oxygen? Participants will be from 2 sub groups:

1. Patients already undergoing TOE (as this is the most common and consistent group who have optiflow- about 4-5 patients per week)
2. Volunteers (staff) who would agree to experience the optiflow whilst awake for the same period as those undergoing TOE

The study will involve a 7 day follow up survey to see if they had experienced complications (runny nose, nasal discomfort, sore throat, epistaxis), what their severity was and how long they lasted for.

ELIGIBILITY:
Inclusion criteria:

1. Volunteers (staff) - from the anaesthetics department and willing to be exposed to HFNO
2. Patients listed for all those undergoing elective TOE requiring sedation and use of HFNO
3. present at Torbay Hospital
4. Greater than 18 years of age. No upper age limit
5. Able to give informed consent

Exclusion Criteria:

1. patient refusal
2. lack of capacity
3. poor understanding of English
4. respiratory tract symptoms
5. blocked nostrils
6. current or recurrent epistaxis
7. nasal steroid treatment
8. Ages <18 years
9. Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory tract symptoms | 7 days
  telephone survey after 7 days

SECONDARY OUTCOMES:
severity of respiratory tract symptoms | 7 days
  telephone survey after 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Katie Flowers, Dr, Principal Investigator — Torbay and South Devon NHS Foundation Trust
Locations (1):
- Torbay Hospital, Torquay, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No